CLINICAL TRIAL: NCT06932094
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of QLS5132 Monotherapy in Subjects With Advanced Solid Tumors
Brief Title: Phase 1 Clinical Study of QLS5132 Monotherapy in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS5132-101
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Finding and Expansion- QLS5132 Monotherapy (Experimental): Intravenous infusion，Q3W
  Interventions: Drug: QLS5132

INTERVENTIONS:
Drug: QLS5132 — antibody drug conjugate (ADC).

SUMMARY:
The Phase 1 trial includes Phase 1a (dose-escalation) and Phase 1b (dose-expansion):

* Phase 1a: Assesses safety, tolerability, PK, and preliminary efficacy of QLS5132 in advanced solid tumors using ATD + BOIN, given IV every 3 weeks. Up to 12 subjects may be enrolled in promising dose levels.
* Phase 1b: Evaluates QLS5132's anti-tumor efficacy in specific CLDN6-positive solid tumors, including ovarian cancer, NSCLC, gastric cancer, and others. Expansion studies at 1~3 selected dose levels follow successful Phase 1a results.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors;
* Measurable disease, per RECIST v1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* Adequate organ function;
* Recover from all reversible AEs from previous anti-tumor treatment (i.e., Grade ≤ 1, according to NCI-CTCAE v5.0), excluding alopecia (any grade) and Grade ≤ 2 neuropathy peripheral;

Exclusion Criteria:

* Previous treatment with drugs targeting CLDN6 (including ADCs), or any drug containing topoisomerase I inhibitors (including ADCs);
* Received prior chemotherapeutic, investigational, or other therapies for the treatment of cancer within 2 weeks with small molecule and within 4 weeks with biologic before the first dose of QLS5132;
* Progressive or symptomatic brain metastases;
* Serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection;
* History of significant cardiac disease, or poorly controlled diabetes mellitus;
* History of recurrent autoimmune diseases;
* History of myelodysplastic syndrome (MDS) or AML;
* History of other active malignant tumors within 3 years before signing the informed consent form;
* If female, is pregnant or breastfeeding;
* Be allergic to any component of QLS5132 or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events | up to 2 years
  Incidence and severity of adverse events, serious adverse events, according to NCI-CTCAE Version 5.0
Maximum tolerated dose (MTD) | 28days
  Highest administered dose with < 33% participants experiencing dose limiting toxicity (DLT) in the first 6 DLT evaluable participants
Recommended Phase 2 Dose (RP2D) | up to 2 years
  Based on the maximum tolerated dose, cumulative safety, and pharmacokinetic data

SECONDARY OUTCOMES:
Maximum Serum Concentration of QLS5132 (Cmax) | 21 days
  PK assessment
Maximum Serum Concentration of QLS5132 at Steady State (Cmax,ss) | 63 days
  PK assessment
Minimum Serum Concentration of QLS5132 at Steady State (Cmin,ss) | 63 days
  PK assessment
Time of Maximum Serum Concentration of QLS5132 (Tmax) | 21 days
  PK assessment
Terminal Half-life (T1/2) of Serum QLS5132 | 63 days
  PK assessment
Area under the Serum Concentration-Time curve from the time of dosing to the last measurable concentration (AUC0-t) for QLS5132 | 21 days
  PK assessment
Area under the Serum Concentration-Time curve from the time of dosing extrapolated to time infinity (AUC0-∞) for QLS5132 | 63 days
  PK assessment
Volume of Distribution (Vd) of QLS5132 | 63 days
  PK assessment
Clearance (CL) of QLS5132 | 63 days
  PK assessment
Objective Response Rate (ORR) | up to 2 years
  Percentage of participants with best response of complete response (CR) or partial response (PR) according to RECIST 1.1
Duration of Response (DOR) | up to 2 years
  Time from CR or PR to objective disease progression or death to any cause
Progression Free Survival (PFS) | up to 2 years
  PFS is defined as the time from the start of the treatment until objective disease progression or death from any cause
Time to Progression (TTP) | 1 years
  Time from start of treatment to disease progression
1 Year Overall Survival (1YOS) | up to 2 years
  Proportion of participants alive at 1 year from the start of treatment to death from any cause
2 Year Overall Survival (2YOS) | 2 years
  Proportion of participants alive at 2 years from the start of treatment to death from any cause
Number of anti-drug antibody (ADA) Positive Participants | up to 2 years
  Immunogenicity will be measured by the number of participants that are ADA positive
Number of neutralizing antibody (Nab) Positive Participants | up to 2 years
  Immunogenicity will be measured by the number of participants that are Nab positive

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, China